CLINICAL TRIAL: NCT02984254
Title: Bracing for Patellofemoral Osteoarthritis. A Prospective Randomized Study of the Treatment of Patellofemoral Arthritis by an Orthosis
Brief Title: Bracing for Patellofemoral Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, MD; PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15016/16
Record Dates: First submitted 2016-10-31; First posted 2016-12-06 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis; Metabolic Disease
Keywords: knee; knee osteoarthritis; Bracing; patellofemoral osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Metabolic Diseases | interventions — Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- functional patellofemoral neoprene brace (Experimental): 26 Patients will use a a functional patellofemoral neoprene brace and answer WOMAC, Lequesne questionnaires, perform Timed-up-and-go (TUG), five-times-sit-to-stand-test (FTSST) and the six-minute walk test.
  Interventions: Device: Womac; Device: Lequesne; Device: Timed-up-and-go (TUG); Device: five-times-sit-to-stand-test (FTSST); Device: Six-minute walk test.; Device: functional patellofemoral neoprene brace
- neoprene sleeve brace. (Experimental): 26 Patients will use a neoprene sleeve brace and answer WOMAC, Lequesne questionnaires, perform Timed-up-and-go (TUG), five-times-sit-to-stand-test (FTSST) and the six-minute walk test.
  Interventions: Device: Womac; Device: Lequesne; Device: Timed-up-and-go (TUG); Device: five-times-sit-to-stand-test (FTSST); Device: Six-minute walk test.; Device: neoprene sleeve brace.

INTERVENTIONS:
Device: Womac — Answer Womac questionnaires at baseline, 1 month, 3 months and 1 year
Device: Lequesne — Answer Lequesne questionnaires at baseline, 1 month, 3 months and 1 year
Device: Timed-up-and-go (TUG) — Perform Timed-up-and-go (TUG) at baseline, 1 month, 3 months and 1 year
Device: five-times-sit-to-stand-test (FTSST) — Perform the five-times-sit-to-stand-test (FTSST) at baseline, 1 month, 3 months and 1 year
Device: Six-minute walk test. — Perform six-minute walk test at baseline, 3 months and 1 year
Device: functional patellofemoral neoprene brace — Use the functional patellofemoral neoprene brace for 2 hours/day minimum - 12 hours/day maximum
  Arms: functional patellofemoral neoprene brace
Device: neoprene sleeve brace. — Use the neoprene sleeve brace for 2 hours/day minimum - 12 hours/day maximum
  Arms: neoprene sleeve brace.

SUMMARY:
BACKGROUND: Despite the prevalence of patellofemoral ostearthritis (OA), this joint has received relatively little attention in the OA literature and there are few treatment options for individuals with patellofemoral OA. Patellar misalignment is associated with radiographic progression patellofemoral OA and symptoms and in magnetic resonance imaging (MRI), to cartilage loss measurements and bone marrow lesions. The hypothesis is that the correction of the patella disorder using strategies such as bracing or adhesive bandages can handle the symptoms and progression of OA.

OBJECTIVE: To compare the effect of a brace designed to stabilize the patellofemoral joint compared with a neoprene sleeve with kneecap opening in patients with patellofemoral OA.

METHODS: Fifty-two patients with patellofemoral OA and co-morbidities (Two or more of: overweight or obesity, hyperglycemia, dyslipidemia, hyperuricemia, high blood pressure) will be divided into two groups according to the knee brace that will receive: Functional Bracing patellofemoral (group 1) and neoprene knee sleeve with patella opening (group 2). Both groups will be oriented on the clinical treatment of osteoarthritis and metabolic syndrome and asked to do daily exercises in addition to reporting the daily consumption of drugs a month before placing the orthotics up to three months after placing it. They will be evaluated with the questionnaires WOMAC and Lequesne, and asked to perform the five-times-sit-to-stand-test, Timed-up-and-go (TUG) and the six-minute walk test in the moments immediately prior to placement of the brace, with one, three and after 12 months bracing.

DETAILED DESCRIPTION:
All patients that sign the informed consent will be randomized and asked to participate in a 4-hour course about knee osteoarthritis. They will be sent home with a form to fill in all medications consumed daily for a month. They will return to the hospital where according to data given by www.randomization.com, they will receive one of two braces in one or both knees depending on their symptoms.

The functional brace has medial, lateral, superior and inferior "ruber bands" that should center patella in the patella groove. The other traditional neoprene sleeve brace with a patellar opening also tries to do the same with no other reinforcement other than the neoprene sleeve.

Prior to bracing, patients will deliver the prior month medication form, answer WOMAC and Lequesne questionnaires, and perform TUG, FTSST and the six-minute walk test.

They will be instructed to use the brace for 2 hours in the first day increasing half an hour per day up to a maximum of 12 hours/day. In case of difficulties with the brace for 12 continuous hours, they will be allowed to use it for at least 4 hours with a 2 hours interval and then again returning to bracing. Patients should sleep/rest without the brace(s). They should use their braces during physical activities unless if under water.

The primary objective is to evaluate and compare the short-term benefits of knee stabilization and compression. Therefore, the follow-up assessments, will be made prior to bracing and after one and three months. The evaluation will include the delivery of the registration of medications consumed daily (along with the hours of use of the orthosis), the WOMAC and Lequesne questionnaires and functional evaluations. X-rays without the braces (Front Schuss, profile and Axial) for measurement of affected joint spaces will be made before inclusion and after one year. Panoramic X-rays of the lower limbs will be performed before inclusion to measure the internal and external femoral-tibial angle. Complaints (pain, slip, swelling, skin lesions) and satisfaction (decrease pain, mobility improvement) with the use of the brace will be sought at each encounter. Patients will be asked about their weekly physical activity (intensity, type and hours of physical activity) on any adverse effects when using orthotics. Weight and height will be measured and each assessment to calculate BMI.

The secondary objective is the improvement in pain, stiffness and long-term function (1 year). Therefore, after a brief analysis of the results of three months, if there is a clinically significant difference between the groups, all patients will use the brace with best results. Therefore the study will be a case series. If both groups show clinically relevant improvements with no significant differences between the orthotics, the study will remain with two arms and the same clinical assessments, questionnaires, functional and radiographic one year. If none of the groups show a clinically relevant improvement in three months, the study will be terminated. Adverse effects of the use of orthotics will also be recorded in the one-year visit. All patients will be advised to discontinue use of the braces and telephone to our secretary in case of any adverse effects in the period between the official evaluations for proper conduct.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic knee OA (patellofemoral)
* Exclusion Criteria:
* Not using the brace as requested;
* Study abandonment;
* No adaptation to brace;
* Skin and vascular complications by use of the brace;
* Failure to complete the consumption of drugs between inclusion and bracing;
* Obesity class II, III or morbid;
* Patients who cannot read or understand the informed consent or the WOMAC questionnaire;

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluate improvement in function | baseline and 3 months
  Apply the Lequesne questionnaire

SECONDARY OUTCOMES:
Improvement in pain | baseline, 1 month, 3 months and 1 year
  Apply the WOMAC questionnaire
Improvement in stiffness | baseline, 1 month, 3 months and 1 year
  Apply the WOMAC questionnaire
Improvement in function with the TUG (Timed-Up-and-Go) | baseline, 1 month, 3 months and 1 year
  Apply TUG (Time-up-Go test)
Improvement in function with Five-Times-Sit-To-Stand-Test (FTSST) | baseline, 1 month, 3 months and 1 year
  Apply Five-Times-Sit-To-Stand-Test (FTSST)
Improvement in function with six minute walk test | baseline, 1 month, 3 months and 1 year
  Apply six minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, MD; PhD, Principal Investigator — Department of Orthopedics and Traumatology - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dillon CF, Rasch EK, Gu Q, Hirsch R. Prevalence of knee osteoarthritis in the United States: arthritis data from the Third National Health and Nutrition Examination Survey 1991-94. J Rheumatol. 2006 Nov;33(11):2271-9. Epub 2006 Oct 1. PMID 17013996
- [Background] McAlindon T, Zhang Y, Hannan M, Naimark A, Weissman B, Castelli W, Felson D. Are risk factors for patellofemoral and tibiofemoral knee osteoarthritis different? J Rheumatol. 1996 Feb;23(2):332-7. PMID 8882042
- [Background] Hunter DJ, Zhang YQ, Niu JB, Felson DT, Kwoh K, Newman A, Kritchevsky S, Harris T, Carbone L, Nevitt M. Patella malalignment, pain and patellofemoral progression: the Health ABC Study. Osteoarthritis Cartilage. 2007 Oct;15(10):1120-7. doi: 10.1016/j.joca.2007.03.020. Epub 2007 May 14. PMID 17502158
- [Background] Kalichman L, Zhang Y, Niu J, Goggins J, Gale D, Felson DT, Hunter D. The association between patellar alignment and patellofemoral joint osteoarthritis features--an MRI study. Rheumatology (Oxford). 2007 Aug;46(8):1303-8. doi: 10.1093/rheumatology/kem095. Epub 2007 May 24. PMID 17525117
- [Background] Hinman RS, Bennell KL, Crossley KM, McConnell J. Immediate effects of adhesive tape on pain and disability in individuals with knee osteoarthritis. Rheumatology (Oxford). 2003 Jul;42(7):865-9. doi: 10.1093/rheumatology/keg233. Epub 2003 Mar 31. PMID 12730546
- [Background] Hinman RS, Crossley KM, McConnell J, Bennell KL. Efficacy of knee tape in the management of osteoarthritis of the knee: blinded randomised controlled trial. BMJ. 2003 Jul 19;327(7407):135. doi: 10.1136/bmj.327.7407.135. PMID 12869456
- [Background] Cushnaghan J, McCarthy C, Dieppe P. Taping the patella medially: a new treatment for osteoarthritis of the knee joint? BMJ. 1994 Mar 19;308(6931):753-5. doi: 10.1136/bmj.308.6931.753. PMID 8142829
- [Background] Crossley KM, Marino GP, Macilquham MD, Schache AG, Hinman RS. Can patellar tape reduce the patellar malalignment and pain associated with patellofemoral osteoarthritis? Arthritis Rheum. 2009 Dec 15;61(12):1719-25. doi: 10.1002/art.24872. PMID 19950307
- [Background] McWalter EJ, Hunter DJ, Harvey WF, McCree P, Hirko KA, Felson DT, Wilson DR. The effect of a patellar brace on three-dimensional patellar kinematics in patients with lateral patellofemoral osteoarthritis. Osteoarthritis Cartilage. 2011 Jul;19(7):801-8. doi: 10.1016/j.joca.2011.03.003. Epub 2011 Mar 11. PMID 21397707
- [Background] Hunter DJ, Harvey W, Gross KD, Felson D, McCree P, Li L, Hirko K, Zhang B, Bennell K. A randomized trial of patellofemoral bracing for treatment of patellofemoral osteoarthritis. Osteoarthritis Cartilage. 2011 Jul;19(7):792-800. doi: 10.1016/j.joca.2010.12.010. Epub 2011 Jan 11. PMID 21232620
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of rheumatoid arthritis. Ann Rheum Dis. 1957 Dec;16(4):485-93. doi: 10.1136/ard.16.4.485. No abstract available. PMID 13498603
- [Background] McCarthy EK, Horvat MA, Holtsberg PA, Wisenbaker JM. Repeated chair stands as a measure of lower limb strength in sexagenarian women. J Gerontol A Biol Sci Med Sci. 2004 Nov;59(11):1207-12. doi: 10.1093/gerona/59.11.1207. PMID 15602077
- [Background] Stratford PW, Kennedy DM, Woodhouse LJ. Performance measures provide assessments of pain and function in people with advanced osteoarthritis of the hip or knee. Phys Ther. 2006 Nov;86(11):1489-96. doi: 10.2522/ptj.20060002. PMID 17079748
- [Background] de Campos GC, Rezende MU, Pailo AF, Frucchi R, Camargo OP. Adding triamcinolone improves viscosupplementation: a randomized clinical trial. Clin Orthop Relat Res. 2013 Feb;471(2):613-20. doi: 10.1007/s11999-012-2659-y. Epub 2012 Oct 26. PMID 23100188
- See also: PARQVE - Project Arthritis Recovering Quality of Life by means of Education. Short-term outcome in a randomized clinical trial — https://www.omicsonline.org/peer-reviewed/parqveproject-arthritis-recovering-quality-of-life-by-means-of-education-shortterm-outcome-in-a-randomized-clinical-trial-20432.html
- See also: . Analysis of anthropometric measures and dietary intake in patients undergoing a multi-professional osteoarthritis education program (PARQVE - Project Arthritis Recovering Quality of Life by means of Education — http://file.scirp.org/pdf/OJO_2016022614241788.pdf
- See also: Translation and cultural validation of the Lequesne's algofunctional questionnaire for osteoarthritis of knee and hip for portuguese language — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0482-50042006000400004